CLINICAL TRIAL: NCT02805114
Title: Obstructive Airways Diseases in Pulmonary Clinic (OADPC) Study
Status: Completed | Type: Observational
Sponsor: Oridion (Industry)
Collaborators: Rabin Medical Center (Other)
Responsible Party: Sponsor
Organization: Medtronic - MITG (Industry)
Other Study IDs: MDT17072
Record Dates: First submitted 2016-06-15; First posted 2016-06-17 (Estimated); Last update posted 2019-01-10 (Actual); Status verified 2019-01

CONDITIONS: Asthma; Chronic Obstructive Pulmonary Disease (COPD)
Keywords: Asthma; Chronic Obstructive Pulmonary Disease (COPD); Capnography
MeSH Terms: conditions — Asthma; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Asthma and COPD patients: Patients with COPD and Asthma. Continuous capnography and spirometry measurements of the subjects will be taken from the subjects with at least two minutes recording before the first spirometry assessment.
  All clinical diagnoses and treatments will be performed according to the department's protocols.
  This is an observational study with no interventions

SUMMARY:
This is an observational study which aims to evaluate the possibility of using data from a capnography device to assess obstructive airway severity in both Chronic Obstructive Pulmonary Disease (COPD) and Asthma patients.

DETAILED DESCRIPTION:
This is an observational study which aims to evaluate the possibility of using data from a capnography device to assess obstructive airway severity in both COPD and Asthma patients. The study will include adult asthma and COPD patients (age >18). Patients will be enrolled on a continuous basis and will be monitored by capnograph and oximeter before and after lung function assessment and also during and after medical treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Age >18
2. Ability and willingness to participate the study and sign informed consent form
3. Asthma / COPD patients

Exclusion Criteria:

1. Pregnant women
2. Asthma or COPD patients with FEV1 > 80%
3. Disability or unwillingness to undergo capnography measurement
4. Cannot be assessed for FEV1
5. Oxygen supply >5 L/min
6. 6. Subjects that gone through LOBECTOMY OF LUNG in the last 5 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Asthma and COPD patients
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2018-05-21 (Actual); Study Completion 2018-05-21 (Actual)

PRIMARY OUTCOMES:
Correlation between capnography parameters and severity of asthma | 1/2 hour to 48 hours from enrollment of subjects
  Correlation between the airway obstruction severity calculation based on the capnography parameters and the clinical severity of asthma and COPD as defined by forced expiratory volume in 1 second (FEV1), in severe asthma and COPD patients

CONTACTS AND LOCATIONS:
Overall Officials: Mordechai M Kremer, Prof.; M.D, Principal Investigator — Rabin Medical Center
Locations (1):
- Pulmonary Institute Rabin Medical center, Beilinson Hospital, Petah Tikva, Israel

IPD SHARING:
Plan to Share IPD: No
Study publication will not contain any identifying data of individuals.

REFERENCES:
- [Derived] Pertzov B, Ronen M, Rosengarten D, Shitenberg D, Heching M, Shostak Y, Kramer MR. Use of capnography for prediction of obstruction severity in non-intubated COPD and asthma patients. Respir Res. 2021 May 21;22(1):154. doi: 10.1186/s12931-021-01747-3. PMID 34020637